CLINICAL TRIAL: NCT02212041
Title: Acceptability, Patterns of Use and Safety of Electronic Cigarette in People With Mental Illness: a Pilot Study
Brief Title: Electronic Cigarettes in Smokers With Mental Illness
Acronym: APUS e-Cigs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 149240
Record Dates: First submitted 2014-08-06; First posted 2014-08-08 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2015-08

CONDITIONS: Schizophrenia; Schizophreniform Disorder; Bipolar Disorder
Keywords: electronic cigarettes; smoking; schizophrenia; serious mental illness
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder; Vaping; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Electronic cigarettes (Experimental): Free disposable electronic cigarettes will be provided during 6 weeks to smokers with serious mental illness.
  Interventions: Other: disposable electronic cigarettes

INTERVENTIONS:
Other: disposable electronic cigarettes — Participants will receive e-cigs free of charge during 6-week. Each week for 6 weeks, participants will receive enough e-cigs to cover 150% of their usual weekly cigarette smoking rate. We will encourage participants to use the e-cigs whenever they would usually smoke a cigarette.
  During a 4-week post-distribution period, we will assess e-cig and cigarette use and other measures when e-cigs are not being freely provided and participants must purchase them on their own. The Week 10 session at the end of this period includes assessment of total nicotine intake, nicotine dependence, subjective and reinforcing effects of e-cigs and cigarettes, attitudes toward e-cigs, motivation to quit and self-efficacy for smoking cessation. At the Week 24 follow-up session we will again collect these measures to determine if any changes observed during the intervention phases have been maintained.
  Other Names: NJOY

SUMMARY:
People with mental illness are more likely to smoke and are more severely addicted to nicotine than the general population. As a result, the number of deaths related to tobacco is higher.

Smoking is highly addictive because it delivers nicotine very quickly. Research studies show that people who use nicotine replacement therapies (such us patches, gums, etc) are more likely to quit smoking than those who try to quit without using these nicotine products. Recently a new electronic nicotine delivery system (ENDS), also known as electronic cigarette (e-cigarette) is rapidly gaining popularity. Electronic cigarettes are devices that mimic traditional cigarettes and deliver nicotine but do not carry the dangerous chemicals contained in tobacco cigarettes.

Given the increasing popularity of e-cigs, there is an urgent need to improve our understanding of both the potential benefits and risks of e-cigs use in people with serious mental illness. In this pilot we propose inviting 50 people with schizophrenia (or schizophrenia-related disorder) who are not intending to quit smoking in the near future to take part in a study in which we will provide 6-weeks of free e-cigs, followed by a 4-week period in which they will not receive free e-cigs and we monitor which products participants choose, and a final 24-week follow-up visit. During the 24-week study period we will assess the use of e-cigs and tobacco cigarettes, the exposure to nicotine and tobacco toxicants, nicotine withdrawal symptoms, the changes in respiratory symptoms and psychiatric symptoms as well as the e-cigs perceived benefits and risks.

ELIGIBILITY:
Inclusion Criteria:

* smokers (≥ 5 cigarettes/day for > 1 yr and breath CO > 5 ppm)
* ages 18-65 years
* ICD-10 diagnosis of schizophreniform, schizophrenia, schizoaffective or bipolar disorder

Exclusion Criteria:

* used e-cigs on > 2 occasions in the past 30 days;
* intend to quit smoking within the next 30 days;
* currently use medications that may reduce smoking (bupropion, varenicline, NRT, naltrexone, buprenorphine, acamprosate, baclofen, clonidine, nortriptyline, anti-seizure medications, disulfiram);
* have unstable psychiatric conditions (hospitalization or change in dose of chronic medication in the past 30 days);
* People with a serious medical condition including uncontrolled high blood pressure, something wrong with their heart or blood vessels that occurred or got worse in the past 3 months (including fast or irregular heart rhythm, angina, chest pain, had a heart attack or stroke).
* People who have ever had a serious stomach ulcer, and/or phaeochromocytoma (tumor of the adrenal gland).
* People who in the last 3 months have had severe heartburn; or a stroke, or unstable kidney disease, unstable liver disease, uncontrolled over-active thyroid gland
* met DSM-IV criteria for drug dependence
* have medical contraindications to nicotine, since nicotine intake may increase in this study;
* have past-month suicidal ideation or past-year suicide attempt.
* are pregnant, as determined through a pregnancy test

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-09-24 (Actual); Primary Completion 2017-05-02 (Actual); Study Completion 2017-05-02 (Actual)

PRIMARY OUTCOMES:
Electronic cigarette use | weekly measurements from baseline to 10 weeks and a final assessment at 24 weeks
  Time Line Follow Back (TLFB) questionnaire
electronic cigarette acceptability | Baseline, week 2, week6, week 10 and week 24
  electronic cigarette evaluation scale (it measures product liking, satisfaction, sensory and physical effects)
Respiratory symptoms | weekly measures from baseline to 10 weeks and at 24 weeks
  An abbreviated and adapted version of the American Thoracic Society Questionnaire (ATS) will be used to assess respiratory symptoms.
Cotinine | Baseline, week 2, 6, 10 and 24
  Cotinine levels in urine
Nitrosamines | Baseline and at 6 week
  NNAL and 3-HPMA levels in urine
Side effects of antipsychotics | weekly the first 10 weeks and at 24 weeks
  The Udvalg for Kliniske Undersøgelser (UKU) scale
Withdrawal symptoms | weekly the first 10 weeks and at 24 weeks
  Mood and Physical Symptoms Scale, MPSS
Respiratory symptoms | weekly the first 10 weeks and at 24 weeks
  Peak Expiratory Flow Rate (PEFR) to monitor airway obstruction, assess its severity and variation.

SECONDARY OUTCOMES:
Predictors of e-Cigs use | Baseline, week 2, 6, 10 and 24.
  Motivation To Stop Scale -MTSS-
Predictors of e-Cigs use | Baseline, week 2, 6, 10 and 24
  Smoking Consequences Questionnaire
Psychiatric symptoms | weekly during the first 10 weeks and at 24 weeks
  Positive and Negative Syndrome Scale
Psychiatric symptoms | weekly the first 10 weeks and at 24 weeks
  Calgary Depression Scale for Schizophrenia
Physical symptoms | weekly the first 10 weeks and at 24 weeks
  Blood pressure and heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Rocio Perez-Iglesias, MD, PhD, Principal Investigator — King's College London; Ann McNeill, BSc, PhD, Prof, Principal Investigator — King's College London; Lynne Dawkins, BSc, PhD, Principal Investigator — University of East London; John Moxham, MD, PhD, Prof, Principal Investigator — King's College London; Philip McGuire, MD, PhD, Prof, Principal Investigator — King's College London
Locations (1):
- South London and Maudsley Foundation Trust (SLaM), London, United Kingdom

REFERENCES:
- [Derived] Hickling LM, Perez-Iglesias R, McNeill A, Dawkins L, Moxham J, Ruffell T, Sendt KV, McGuire P. A pre-post pilot study of electronic cigarettes to reduce smoking in people with severe mental illness. Psychol Med. 2019 Apr;49(6):1033-1040. doi: 10.1017/S0033291718001782. Epub 2018 Jul 10. PMID 29986786